CLINICAL TRIAL: NCT02350985
Title: Effectivity of Propranolol and Venlafaxine in Treatment of Vestibular Migraine: A Randomized Controlled Clinical Trial
Brief Title: Comparison of Propranolol and Venlafaxine in Treatment of Vestibular Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehti Salviz, MD, Attending ENT surgeon, Haseki Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HasekiTRH
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Vestibular Migraine
Keywords: Migraine; Migrainous Vertigo; Headache Disorders; Central Nervous System Origin Vertigo; Paroxysmal Vertigo; Adrenergic beta-Antagonist; Vasodilator Agent; Anti Arrhythmia Agent; Serotonin Uptake Inhibitor; Antidepressive Agent; Propranolol; Venlafaxine
MeSH Terms: conditions — Migraine Disorders; Headache Disorders; Vertigo | interventions — Propranolol; Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol (Active Comparator): Propranolol up to 160 mg/day
  Interventions: Drug: Propranolol
- Venlafaxine (Active Comparator): Venlafaxine up to 150 mg/day
  Interventions: Drug: Venlafaxine

INTERVENTIONS:
Drug: Propranolol — Propranolol was given in a flexible dose between 40 mg to 160 mg with an escalating fashion starting at 40 mg PO AM for one week and followed by 40 mg AM and 40 mg PM for a total dose up to 160 mg daily
  Other Names: Dideral
  Arms: Propranolol
Drug: Venlafaxine — Venlafaxine treatment was followed as: 37.5 mg qhs for two weeks and followed 75 mg qhs with an escalating dose with 2 weeks periods up to 150 mg daily
  Other Names: Efexor
  Arms: Venlafaxine

SUMMARY:
The presented study aims to compare effectivity of propranolol with effectivity of venlafaxine in escalating dose in subjects with vestibular migraine (VM) over a period of 12 weeks. The study population consisted of subjects diagnosed definite VM according to criteria of Bárány Society and Migraine Classification Subcommittee of the International Headache Society (IHS). Effectivity of therapy was measured by Dizziness Handicap Inventory (DHI), number of vertiginous attack of last month and visual analogue scale (VAS) reported dizziness related Quality of Life (QOL). Beck Anxiety Inventory (BAI) and Beck Depression Inventory (BDI) were also used to determine psychiatric improvement played role in response to therapy in venlafaxine treatment arm.

DETAILED DESCRIPTION:
Vestibular migraine (VM) is a condition of episodic vertigo linked to migrainous symptoms described by Nueuhauser et al. in 2001. Some subjects benefit behavior and diet modification and controls of their symptoms. Anti-migrainous medication for prophylactic aim is given subjects who do not benefit life-style improvement. However, there is absence of sufficient evidence for treatment of VM.

In this study the investigators aimed to evaluated effectiveness of prophylactic treatment venlafaxine by comparing propranolol in VM. The investigators also aimed to investigate if the effectiveness of venlafaxine is linked to the improvement of psychiatric condition.

All subjects who were suspected to having VM referred to both M.S. (Department of Otolaryngology) and H.A. (Department of Neurology) in order to ensure subjects fill the criteria of VM and did not have other vestibular disorders. All subjects underwent detailed neurologic, neurotologic examination, audiometric investigation, videonystagmography (VNG) and bithermal caloric testing in order to exclude other or additional vestibular or neurologic disease. Subjects who were18 years or old with a history of (at least 2 months) definite VM according to criteria of Bárány Society and Migraine Classification Subcommittee of the International Headache Society (IHS) were eligible for this study. After a subject fill the eligibility criteria of the study who did not respond to lifestyle or dietary modification were enrolled to the study.

Subjects were enrolled to the study if they filled to the inclusion and exclusion criteria and written informed consent was obtained from all subjects. Subjects were randomized using sealed envelop methods by A.K. (Department of Otolaryngology). Before starting intervention protocol Dizziness Handicap Inventory (DHI), number of vertiginous attack of last month and visual analogue scale (VAS) reported dizziness related Quality of Life (QOL), Beck Anxiety Inventory (BAI) and Beck Depression Inventory (BDI) were obtained from all subjects by T.Y. (Department of Otolaryngology). Subjects were given propranolol or venlafaxine treatment according to randomization with balanced allocation (1:1). The study was unblinded because the study is not an investigational and propranolol was paid by government health insurance. However, venlafaxine is not paid for the migraine therapy by government health insurance and venlafaxine was provided by Institution Research Funding System.

The intervention protocol was carried on by T.Y. under supervision of H.A and M.S.. Propranolol was given in a flexible dose between 40 mg to 160 mg with an escalating fashion starting at 40 mg PO AM for one week and followed by 40 mg AM and 40 mg PM for a total dose up to 160 mg daily. Venlafaxine treatment was followed as: 37.5 mg qhs for two weeks and followed 75 mg qhs with an escalating dose with 2 weeks periods up to 150 mg daily. All participants were asked to self-titrate their medication in case if inform the researchers. Subjects were to be seen at the clinic biweekly for first month in order to evaluated adverse effects and to make sure participants were having sufficient dosage. The effective duration of the treatment was considered as 3 months and participants were asked to continue using their medication one more month in order to evaluate change from baseline to 3rd month in terms of number of vertiginous attacks of the last month. All participants were assessed at the clinic at month 1, 3 and 4. Change from baseline DHI, VAS, BAI and BDI were scored at 4th month.

Adverse effects, reason to exclude the subjects from the study, reason subjects refused to continue the study and other reasons subjects could not follow the protocol were all recorded during clinic visits or obtained over the phone at home.

The analysis primary endpoint was performed following the intention-to-treat (ITT) method. Missing data was handled by multiple imputation method.

ELIGIBILITY:
Inclusion Criteria:

* vestibular migraine does not respond lifestyle and dietary modification

Exclusion Criteria:

* known allergic reaction to venlafaxine or propranolol
* under the care of psychiatrist
* pregnancy or intention to become pregnant
* presence significant illness or medical condition such as cancer, liver or kidney failure
* certain medical conditions with possible adverse effects with propranolol or venlafaxine following as: AV block or bradyarrhythmia; astma or COPD; diabetes mellitus.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Dizziness Handicap Inventory | 4 months post randomization

SECONDARY OUTCOMES:
Change from baseline in Beck Anxiety Inventory | 4 months post randomization
Change from baseline in Beck Depression Inventory | 4 moths post randomization
Change from baseline in dizziness related quality of life | 4 moths post randomization
  Dizziness related quality of life score by visual analog scale
Change number of vertiginous attack | 3 moths post randomization
  Baseline of number of attacks were obtained 1 moths before randomization and months between 3 and 4 moths after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)